CLINICAL TRIAL: NCT01901237
Title: Impact of Yoga on Quality of Life for Adolescent and Young Adult Non-Curative Cancer Patients: A Pilot Study
Brief Title: Yoga for Adolescent and Young Adult Non-Curative Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Rutledge (Other)
Collaborators: Dalhousie University (Other); IWK Health Centre (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Rob Rutledge, Associate Professor, Department of Medicine, Dalhousie University, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDHA-RS/2014-067
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Advanced Cancer
Keywords: Cancer; Adolescent and Young Adult; Exercise; Physical Activity; Quality of Life; End-of-Life; Palliative; Terminal; Yoga; Alternative Therapies; Fitness; Fatigue
MeSH Terms: conditions — Neoplasms; Motor Activity; Death; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hatha Yoga Program (Other): Single-arm pilot study of a 7-week home/hospice-based Hatha yoga program for adolescent and young adults with non-curative cancer.
  Interventions: Behavioral: Hatha Yoga

INTERVENTIONS:
Behavioral: Hatha Yoga — This is a 7-week home/hospice-based instructive Hatha yoga program (available on DVD) for adolescent and young adults diagnosed with a non-curative cancer. Participants will be asked to complete a minimum of one, 75-minute yoga session per week. The DVD package includes four discs that increase in difficulty over the course of the 7-week program. The DVD focuses on postures and breathing exercises. Participants will be asked to keep track of the number and duration of yoga sessions completed over the 7-week period.

SUMMARY:
Adolescents and young adults who are living with cancer are not benefiting from the same age-appropriate physical and psychosocial care, as are children and older adults. As a result, their unique needs often go unmet or unaddressed. Studies have demonstrated that a lack of age-appropriate care may be responsible for a deceased quality of life. Studies have also shown that physical activity is able to reduce many of the negative side-effects linked to cancer and its treatment (e.g., nausea, vomiting, fatigue). A light form of physical activity that is both safe and manageable for cancer patients is yoga. The purpose of this study is to examine the achievability and safety of a light 7-week home/hospice-based Hatha yoga program (available on DVD) in the adolescent and young adult non-curative cancer population. This study will also examine the ability of yoga to reduce cancer related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a non-curative cancer and assigned to non-curative or palliative care
* Between 15-39 years of age
* Have primary physician/oncologist consent to participate

Exclusion Criteria:

* Experience any medical conditions that contraindicate yoga (e.g., bone metastases)
* Exhibit cognitive limitations (e.g., psychiatric disorders)
* Score below 30% on Palliative Performance Status Scale

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment | Final: end of week 7
  Recruitment will be calculated by the number of patients who consent to participate, divided by the number of eligible participants recommended by the primary oncologist/physician.
Feasibility: Retention | Final: end of week 7
  Retention: Will be determined by reporting the number of participants who complete the baseline and post-program questionnaire and follow-up testing.
Feasibility: Adherence | Final: end of week 7
  Adherence: Participants will be asked to record the number of yoga sessions performed each week. Overall adherence will be calculated by summing the actual number of sessions the participant engaged in, divided by the recommended number of sessions.
Safety | Final: end of week 7
  Safety: Any adverse events reported by the participant will be recorded.

SECONDARY OUTCOMES:
Changes in Quality of Life | Baseline: week 1; Final: week 7
  Participants will be asked to complete the Functional Assessment of Chronic Illness Therapy - Palliative Care subscale (FACIT-Pal) and the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being subscale (FACIT-Sp) at baseline and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Rutledge, MD, FRCPC, Principal Investigator — Capital District Health Authority, Halifax, Canada
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: Published abstract. — http://ascopubs.org/doi/abs/10.1200/jco.2016.34.3_suppl.249